CLINICAL TRIAL: NCT04739293
Title: Phase 1 Study to Assess the Safety, Tolerability, and Pharmacokinetics of ON 123300 Capsules Administered Orally as Escalating Daily Doses in Patients With Advanced Cancer Relapsed or Refractory to at Least One (1) Prior Line of Therapy
Brief Title: Study of ON 123300 in Patients With Advanced Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Traws Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19-01
Record Dates: First submitted 2021-01-29; First posted 2021-02-04 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Solid Tumors, Adult
MeSH Terms: interventions — ON123300

STUDY DESIGN:
Intervention Model Description: 3+3 dose escalation design with expansion cohort at recommended phase 2 dose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ON 123300 (Experimental): ON 123300 capsules at increasing doses per cohort, starting at 40 mg
  Interventions: Drug: ON123300

INTERVENTIONS:
Drug: ON123300 — ON 123300 hard gelatin capsules
  Other Names: HX 301

SUMMARY:
This study will investigate the safety of the drug ON 123300 at increasing doses to determine the best dose to use in future clinical trials.

DETAILED DESCRIPTION:
After being informed about the study including potential risks, patients giving written informed consent will proceed to a screening period when assessments will be performed to determine whether the patient is eligible to participate in the study. If the patient is eligible, they will start to receive ON 123300 as capsules every day. On day 1 and Day 8 of the study, patients will be required to provide eight blood samples to allow measurement of the amount of drug in their blood. Three ECGs will also be performed during this time. Patients will continue to receive ON 123300 until disease progression, unacceptable toxicity, or patient or physician decision to stop.

The first group of patients will receive 40mg of ON 123300 daily, the next group 80mg of ON 123300, the 120mg, etc. until the correct dose has been determined for future studies.

Patients will visit the clinic on Days 1, 2, 8, and 9, then weekly for the first month, then every two weeks for two more months, then every month.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age the time of signing the informed consent form (ICF);
2. Histological or cytological evidence of advanced and/or metastatic cancer,

   1. For Dose Escalation Cohorts, patients with measurable or non-measurable disease;
   2. For RP2D Expansion Cohort, patients with measurable disease;
3. Patients must have received and failed at least one prior approved treatment, or have no therapeutic options available as deemed appropriate by their treating physician;
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of < 2;
5. Life expectancy of > 3 months;
6. Patients must be able to swallow oral capsules;
7. Women of child-bearing potential must have a negative serum screening for pregnancy within 14 days prior to screening. Women and men of child-bearing potential must agree to use highly effective methods of birth control before entry and throughout the study, for up to 12 weeks following the last dose of ON 123300.
8. Patients must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted;
9. Patients must have the ability to understand the nature of the study and any hazards of participating in the study and communicate satisfactorily with the investigator to participate in the study.
10. Patients must be willing and able to adhere and comply to the requirements of the entire study including study visit schedule and other protocol requirements;
11. Have adequate organ function, including:

    a. Hematologic: i. absolute neutrophil count (ANC) ≥1.0 × 109/Liter (L) ii. platelets ≥100 × 109/L, and iii. hemoglobin ≥8 g/deciliter (dL). b. Hepatic: i. Total bilirubin ≤1.5 times the upper limit of normal (ULN) and ii. alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3.0 times ULN (or ALT and AST ≤5 times ULN if liver metastases are present).

    c. Renal: i. Serum creatinine ≤1.5 times ULN. or estimated creatinine clearance (calculated according to normal institutional practice) greater than 50 ml/min.

Exclusion Criteria:

1. Patients that have any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the patient from participating in the study or present an unacceptable risk to the patient;
2. Patients at risk for Torsades de pointes (TdP):

   1. Who have a marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >480 milliseconds (ms) (CTCAE grade 1) using Fredericia's QT correction formula, or
   2. who have a history of additional risk factors for TdP (e.g., heart failure, hypokalemia, family history of Long QT Syndrome), or
   3. who are currently taking medications that prolong the QT/QTc interval;
3. Patients with a diagnosis of hematological malignancies except for non-Hodgkin's lymphoma;
4. Have received recent chemotherapy, hormonal therapy, other targeted cancer treatment, or investigational therapy within 14 days of planned first dose;
5. Patients currently taking or within 5 half-lives of taking strong inducers and inhibitors of CYP2C8 and CYP3A4;
6. History of allergic reaction attributed to compounds of similar chemical or biologic composition/structure to ON 123300 (e.g. prior CDK4/6 inhibitors);
7. Uncontrolled intercurrent illness including but not limited to ongoing or active infection, bleeding, congestive heart failure, unstable angina, cardiac arrhythmia, oxygen-dependent lung disease, psychiatric illness/social situations that limit participation compliance with study procedures and requirements;
8. Patients with a recent history of venous thromboembolic events, defined as event occurring ≤ 6 months prior to screening and also currently on therapy;
9. Patients with baseline Grade ≥ 2 diarrhea;
10. Patients with Grade ≥ 3 hypercalcemia (Corrected serum calcium > 12.5 mg/dL);
11. Pregnant or nursing mothers;
12. Have had major surgery within 14 days prior to screening to allow for post-operative healing of the surgical wound and site(s).
13. Have received recent (within 28 days prior to screening) live attenuated vaccines.
14. Have active bacterial, fungal or detectable viral infection (e.g. Human Immunodeficiency Virus or Hepatitis B or Hepatitis C).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-05-13 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLT) | First 28 days of dosing
  Incidence of protocol defined toxicities that would result in stopping dosing
Incidence of adverse events (AE) | Consent to 30 days after last dose
  Adverse events as measured by CTCAE version 5.0
Abnormal Laboratory Test results | Consent to 30 days after last dose
  Changes and trends in standard hematology and chemistry blood tests

SECONDARY OUTCOMES:
Establish the recommended phase 2 dose (RP2D) | First 28 day cycle
  Incidence of DLTs
Pharmacokinetics of ON 123300 and 2 metabolites - Cmax | Intense PK on Cycle1 Day1 and Day 8; Single samples pre-dose on Cycle 2 Day 1 and Cycle 3 Day 1 (each cycle is 28 days)
  Maximum plasma concentration
Pharmacokinetics of ON 123300 and 2 metabolites - Tmax | Intense PK on Cycle1 Day1 and Day 8; Single samples pre-dose on Cycle 2 Day 1 and Cycle 3 Day 1 (each cycle is 28 days)
  Time to reach Cmax
Pharmacokinetics of ON 123300 and 2 metabolites - AUClast | Intense PK on Cycle1 Day1 and Day 8; Single samples pre-dose on Cycle 2 Day 1 and Cycle 3 Day 1 (each cycle is 28 days)
  The area under the plasma concentration-time curve (AUC) calculated to the last quantifiable sample
Pharmacokinetics of ON 123300 and 2 metabolites - T1/2 | Intense PK on Cycle1 Day1 and Day 8; Single samples pre-dose on Cycle 2 Day 1 and Cycle 3 Day 1 (each cycle is 28 days)
  Terminal phase elimination half-life
Pharmacokinetics of ON 123300 and 2 metabolites - CL/F | Intense PK on Cycle1 Day1 and Day 8; Single samples pre-dose on Cycle 2 Day 1 and Cycle 3 Day 1 (each cycle is 28 days)
  The apparent oral clearance
Pharmacokinetics of ON 123300 and 2 metabolites - Vss | Intense PK on Cycle1 Day1 and Day 8; Single samples pre-dose on Cycle 2 Day 1 and Cycle 3 Day 1 (each cycle is 28 days)
  Steady state volume of distribution

OTHER OUTCOMES:
Preliminary efficacy of ON 123300 | Through study completion, an average of 6 months
  Objective responses by RECIST

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Saunders, MD, Study Director — Onconova Therapeutics
Locations (3):
- United States (3):
  - START Midwest, Grand Rapids, Michigan
  - Greenville Health System, Institute for Oncology Clinical Research, Greenville, South Carolina
  - Mary Crowley Cancer Research, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No